CLINICAL TRIAL: NCT03802474
Title: Biomechanical Assessment of Spinal Posture in Girls With Primary Dysmenorrhea
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, HAhmed, lecture of biomechanics, Cairo University
Other Study IDs: P.T.REC/012/002074
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2018-09

CONDITIONS: Primary Dysmenorrhea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: girls with primary dysmenorrhea subject to three-dimensional analysis of the back will conducted with the 4D formetric device and inclinometer to measure range of motion of spine
- Group B: girls with normal painless menstruation without primary dysmenorrhea subject to three-dimensional analysis of the back will conducted with the 4D formetric device and inclinometer to measure range of motion of spine

SUMMARY:
Dysmenorrhea comes from the Greek word for difficult monthly flow and describes painful menstruation.Primary dysmenorrhea might be caused by spinal misalignment and incompatibility between muscles of the pelvic circumference and soft tissue.Leg Length Discrepancy affects spinal posture. Although, several studies evaluated the relation between spinal alignment, spinal configuration and primary dysmenorrhea, but, there is no previous study investigate the effect of leg length discrepancy on primary dysmenorrhea. So, this study will correlate leg length discrepancy with spinal configuration and primary dysmenorrhea.

Statement of the problem:

Is there an impact of spinal posture on primary dysmenorrhea in girls?

Hypothesis:

Null hypothesis: There is no impact of spinal mobility ,spinal configurations and leg length discrepancy on primary dysmenorrhea

DETAILED DESCRIPTION:
Primary dysmenorrhea is defined as painful menses in women with a normal pelvic anatomy. Adolescent girls tend to have a higher prevalence of primary dysmenorrhoea than older women, as primary dysmenorrhoea can improve with age.Asymmetry in upright posture is associated with various outcomes, such as the decreased loading of the affected side in stroke; degenerative changes of the hip, knee, and ankle joints and spine; or a leg length discrepancy.restriction of movement of the lumbosacral vertebrae, body fluid increases within the pelvis as well as contraction of the uterus leading to the intensification of the menstrual pain. Although, several studies evaluated the relation between spinal alignment, spinal configuration and primary dysmenorrhea, but, there is no previous study investigate the effect of leg length discrepancy on primary dysmenorrhea. So, this study will correlate leg length discrepancy with spinal configuration and primary dysmenorrhea.

One handred healthy girls with regular menstrual cycle and are not have any pelvic or gynecological disorders will be participated in this study. All subjects will be recruited from student of faculty of physical therapy, Cairo University.

1. Personal data: All data will be recorded in a recording data sheet.
2. Formetric Raster stereography: It will be used to assess spinal configuration (kyphotic angle, lordotic angle, pelvic inclination, trunk inclination and pelvic tilting) during menstruation.
3. Leg length discrepancy Tape measure can be used to measure the true leg length from the anterior superior iliac spine to the medial malleolus. The functional leg length is measured from the umbilicus to medial malleolus.
4. Inclinometer can be used to measure range of motion of lumbar spines.

ELIGIBILITY:
Inclusion Criteria:

* Healthy girls with regular menstrual cycles with an average of 28:35 days.
* Their age will be ranged from 17to 24 years.
* Their body mass index will be ranged from 20 to 25kg/m2.

Exclusion Criteria:

* Girls who have musculoskeletal disorders as low back pain.
* Girls who have any pelvic or gynecological disorders.
* History of lower limb injury.
* Over-weight and obese girls.
* Thin and underweight girls.
* Girls with spinal deformities as kyphosis and scoliosis.

Ages: 17 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — healthy girls with regular menstrual cycle and are not have any pelvic or gynecological disorders will be participated in this study
Study Population: Healthy girls with regular menstrual cycle and are not have any pelvic or gynecological disorders will be participated in this study. All subjects will be recruited from student of faculty of physical therapy, Cairo University.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Trunk inclination | 1month
  the trunk inclination refer to the difference in height between VP and DM based on a vertical plane (sagital section).
  an angle >2.8 referred to as " Inclination" (I), an angle <2.8 as "reclination" (R).
Kyphotic angle | 1 month
  this is the maximum kyphotic angle measured between the surface tangents of the upper inflection point ICT in the vicinity of the VP and the thoracic lumbar inflection point ITL.
lateral deviation | 1 month
  the total deviation of the spinal midline from the VP-DM line in the frontal plane , i.e the maximum deflection on the right plus the maximum deflection on the left
lordotic angle | 1 month
  this is the maximum lordotic angle measured between the surface tangents of the thoracic-lumbar inflection point ITL and the lower lumbar-sacral inflection point ILS
pelvic inclination | 1 month
  this is calculated as the mean torsion of the DLand DR surface normals
pelvic tilt | 1 month
  the difference in height of the lumbar dimples, based on a horizontal plane (transverse section ). DR is higher than DL if the angle is positive
pelvic torsion | 1 month
  pelvic torsion is calculated from the reciprocal torsion of the surface normals on the two lumbar dimples (vertical components). If the difference angle is positive, then the normal on the right dimple (DR) is up more than on the left dimple.

SECONDARY OUTCOMES:
leg lenght discripancy | 1 months
  True leg length is measured from the anterior superior iliac spine to the medial malleolus. The functional leg length is measured from the umbilicus to medial malleolus.

OTHER OUTCOMES:
Trunk flexion | 1 month
  Flexion describes a bending movement that decreases the angle between a segment and its proximal segment
Trunk extention | 1 month
  Extention describes a straightening movement that increases the angle between body parts
trunk lateral flexion | 1 month
  Lateral flexion describes bending movement of a body part in the lateral direction, that is to say sidewards. It can be performed either to the right or to the left side.